CLINICAL TRIAL: NCT05743699
Title: Adaptation and Evaluation of Bright Horizons: An Evidence Based Intervention for Prevention of Binge Drinking and Drug Use
Brief Title: Adaptation and Evaluation of Bright Horizons
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Native American Research Center for Health (Other); White Mountain Apache Tribe (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00021437
Record Dates: First submitted 2023-02-15; First posted 2023-02-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Abuse; Substance Use
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case management + Bright Horizons (Experimental): Participants enrolled into the Bright Horizons intervention group will receive one 2-4 hour long session with an Research Program Assistant.
  Interventions: Behavioral: Bright Horizons; Behavioral: Case Management
- Case management (Placebo Comparator): Participants in the control group will receive standard case management via the White Mountain Apache suicide and self-harm surveillance system.
  Interventions: Behavioral: Case Management

INTERVENTIONS:
Behavioral: Bright Horizons — Bright Horizons is a brief substance use intervention delivered by Research Program Assistants.
  Arms: Case management + Bright Horizons
Behavioral: Case Management — Placebo condition

SUMMARY:
This study will test if a program called 'Bright Horizons' is effective at reducing binge substance use among adolescents.

Bright Horizons is a culturally adapted intervention developed and tested through a partnership between The White Mountain Apache Tribe and Johns Hopkins University. Bright Horizons is a brief intervention that teaches emotion regulation, coping skills, and problem solving. The intervention also uses goal setting to reduce alcohol and other substance use and to connect to individuals with treatment.

DETAILED DESCRIPTION:
The goal of this study is to understand how Bright Horizons impacts adolescents who have a recent binge substance use event. Participants will receive a lesson on binge substance use and answer questions at three different time points: when participants enroll in the study; 4 weeks later; and 4 weeks after that visit. Evaluation questions will ask about participants' substance use, family and peer relationships, and other emotions and behaviors.

Control participants will receive the Bright Horizons intervention after enrollment of all intervention participants is complete.

ELIGIBILITY:
Inclusion Criteria:

* Aged 12-17
* Confirmed binge alcohol use event reported to the surveillance system within 90 days
* Self identify as Native American
* Reside on or near the Fort Apache Indian Reservation
* Have parental or legal guardian consent/provide youth assent

Exclusion Criteria:

* Unstable and severe medical, psychiatric or drug use problems that necessitates inpatient treatment
* Acute suicidal or homicidal ideation requiring immediate intervention
* Recent and severe stressful life events such as physical or sexual abuse, or violent crime victimization that requires specific and high intensity interventions or out of home placement
* Doesn't speak English
* Severally visually impaired

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Alcohol Use as assessed by Timeline Followback | Baseline, 4 weeks and 8 weeks post-intervention
  Alcohol use over the past 30 days (Timeline Followback to assess number of drinking days and number of drinks per day)

SECONDARY OUTCOMES:
Coping with Stressful Life Events as assessed by the Difficulties in emotion regulation scale | Baseline, 4 weeks, and 8 weeks
  Difficulties in emotion regulation scale is a 36-item instrument that asks individuals to rate their difficulties in regulating emotions including non-acceptance of emotional responses, awareness of emotions and access to regulation strategies. Scores can range from 36 to 180, with higher scores indicating more difficulties in regulating emotions.
Impulsivity as assessed by the UPPS Impulsive Behavior Scale | Baseline, 4 weeks, 8 weeks
  UPPS Impulsive Behavior Scale is a 45-item inventory designed to measure four personality pathways to impulsive behavior: Urgency to Act, Lack of Perseverance, Lack of Premeditation, and Sensation Seeking, each rated on a 4-point scale. Scores can range from 45 to 180, with higher scores indicating more impulsivity.
Family Functioning as assessed by the Problem-oriented screening instrument (POSIT) Family Functioning scale | Baseline, 4 weeks, 8 weeks
  Problem-oriented screening instrument (POSIT) Family Functioning Items is a 10 item scale that measures family functioning around parenting, communication and child monitoring. Responses No=0 and Yes=1. A score of 8 shows healthier family functioning, and a score of 2 shows worse family functioning.
Peer Relationships as assessed by the Peer Norms questionnaire | Baseline, 4 weeks, 8 weeks
  Peer Norms measure is a 20-item measure asking about peer behaviors and the participant's perception of peer behaviors. Topics include sexual activity, drinking and other substance use. Peer groups discussed include best friends, people in their grade, and people their age. Scores can range from 11 to 60, with higher scores indicating more peer pressure and less healthy peer relationships.
Other substance use as assessed by the Youth Risk Behavior Survey (YBBS) | Baseline, 4 weeks, 8 weeks
  Youth Risk Behavior Survey (YRBS) was developed so youth can describe their behaviors that may affect their health. For this study, 19 items have been selected that ask about alcohol, marijuana, and other substance use. Scores can range from 0 to 99, with higher scores indicating more/worse substance use.
Enculturation as assessed by the Tribal identification scale | Baseline, 4 weeks, 8 weeks
  Tribal identification scale comprises 7 questions that ask about identity and connection to ones tribal community. Scores can range from 7 to 35, with higher scores indicating less connection with tribal community.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Cwik, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Center for Indigenous Health - Whiteriver Site, Whiteriver, Arizona, United States

IPD SHARING:
Plan to Share IPD: No